CLINICAL TRIAL: NCT07063251
Title: An Investigator-initiated, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of HG005 in Pediatric Patients With Stargardt Disease (STGD1) Caused by Biallelic ABCA4 Mutations
Brief Title: An Clinical Study Evaluating the Safety, Tolerability, and efficAcy of HG005 in StaRgardT Disease
Acronym: START
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: HuidaGene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG00501
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Stargardt Disease Type 1 (STGD1)
Keywords: Stargardt disease type 1 (STGD1); Stargardt Macular Dystrophy; Stargardt Macular Degeneration; HG005; AAV; Gene Therapy
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HG005 (Experimental): The study will enroll up to 2 dose cohorts
  Interventions: Genetic: HG005

INTERVENTIONS:
Genetic: HG005 — Once subretinal injection; The duration of the study is about 52 weeks for each subject, including a 4 weeks screening period, enrollment visit, treatment visit, and 56 weeks follow-up period.

SUMMARY:
Stargardt disease type 1 (STGD1) is a rare genetic eye condition that causes progressive vision loss, often beginning in childhood or adolescence. It is the most common form of inherited macular degeneration and can lead to legal blindness. STGD1 is caused by mutations in the ABCA4 gene, which normally helps clear waste from the photoreceptor cells in the retina. When ABCA4 gene doesn't function properly, toxic substances like A2E accumulate and damage the retinal pigment epithelium (RPE), leading to vision loss.

There are currently no approved treatments for STGD1. HG005 is an investigational gene therapy designed to deliver a healthy copy of the ABCA4 gene to the retina. Because the gene is too large to fit into a single AAV (adeno-associated virus) vector, HG005 used two AAV vectors that work together in retinal cells to produce the full-length, functional ABCA4 protein. The goal of HG005 is to restore normal waste removal, protect retinal cells from further damage, and slow or stop vision loss.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 6 and ≤17 years at the time of signing informed consent, with clinical diagnosis of Stargardt disease;
* At least one ABCA4 allele on each chromosome;
* Both eyes must have well-defined macular atrophic lesions consistent with the diagnosis of Stargardt macular dystrophy.
* Meet visual acuity criteria based on ETDRS letter chart
* Subject must agree to contraception during the study.
* Acceptable hematology, clinical chemistry, urine laboratory, and protocol required eye examination.

Exclusion Criteria:

* Presence of active intraocular inflammation or uveitis history in either eye;
* Presence of ocular or periocular infection history in either eye within 2 weeks prior to selection;
* History or presence of corneal dystrophy in the study eye;
* History of HIV or hepatitis A, B, or C infection;
* Previous treatment with any gene therapy or cell therapy (e.g., stem cell transplantation);
* Additional intraocular surgery in study eye 3 months prior to baseline visit;
* Participation in an oral therapeutic STGD clinical trial within 3 months (or within 5 half-lives after last dose) prior to Screening
* Any concomitant treatment that, in the opinion of the investigator, might interfere with the surgical procedure or healing process of the eye
* Any other conditions that would not allow the potential subject to complete follow-up examinations during the study and would, in the opinion of the investigator, make the potential subject unsuitable for the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of systemic adverse events | 26 & 52 weeks
  Number of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Change of study eye versus control eye in Low Luminance Visual Acuity(LLVA) | 52 weeks
Change of study eye versus control eye in Fundus Autofluorescence (FAF) | 52 weeks
Change of study eye versus control eye in Optical Coherence Tomography (OCT) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — HuidaGene Therapeutics Co., Ltd.
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China